CLINICAL TRIAL: NCT03591263
Title: Longitudinal Study of Clinical Outcomes in Patients Referred to Pulmonary Rehabilitation
Brief Title: Clinical Outcomes in Patients Referred to Pulmonary Rehabilitation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805017RINB
Record Dates: First submitted 2018-06-12; First posted 2018-07-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic obstructive pulmonary disease: Subjects with the diagnosis of chronic respiratory disease, such as chronic obstructive pulmonary disease, bronchiectasis, idiopathic pulmonary fibrosis that referred for evaluation as routine care at Physical Therapy Center (National Taiwan University)
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pulmonary rehabilitation as routine care includes, airway clearance techniques, breathing exercise, and physical training instruction

SUMMARY:
Chronic obstructive pulmonary disease is a chronic inflammatory lung disease that causes obstructed airflow from the lung, characterized by chronic cough, dyspnea, and sputum production, which often misunderstood as aging or catching a cold. These symptoms may be progressive over time. To provide better disease management and early detecting, pulmonary rehabilitation is now considered a fundamental component of the integrated disease management of this population. However, few studies have evaluated the beneficial outcomes in patients referred to pulmonary rehabilitation. Therefore, the purpose of this study is to investigate the clinical outcomes in patients referred to pulmonary rehabilitation in National Taiwan University Hospital.

ELIGIBILITY:
Inclusion criteria:

1. age > 20 years old
2. patients with chronic respiratory disease diagnosed by physician that referred to pulmonary rehabilitation in National Taiwan University Hospital including, chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, bronchiectasis
3. can cooperate with pulmonary rehabilitation clinic

Exclusion criteria:

1. angina, acute myocardial infarction in the previous one month
2. pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic respiratory disease: chronic obstructive pulmonary disease, idiopathic pulmonary fibrosis, bronchiectasis.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-06-25 (Actual); Primary Completion 2024-06-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity using the six-minute walk test | The six-minute walk test needs six minute to complete the test
  The six-minute walk test is commonly performed to evaluate functional exercise capacity. The six-minute walk test was performed according to the guidelines, and the distance walked in the test presented as functional exercise capacity.
Muscle strength: hand grip | Hand grip of both hands need about three minutes to complete
  Hand grip strength is performed by using hand dynamometer
Lung hygiene | Lung hygiene is evaluated as the frequency of acute exacerbation in the the past one year
  Lung hygiene is evaluated by the frequency of acute exacerbation
Home-based physical activity | Record the home-based physical activities everyday that the subjects have in the past one week that lasting for one year.
  All subjects were encouraged to increase their daily physical activity and recorded the amount of physical activity on patient-self-record training log.
Muscle strength: leg press | Maximum leg press measurement needs about four minutes to complete
  Maximum leg press is performed by using seated leg press machine
Heart rate | Hospital-based physical training takes 30 minutes, once a week, and it also takes 30 min to measure continuously
  Heart rate is measured at rest, during hospital-based physical training.
Blood pressure | Hospital-based physical training takes 30 minutes, once a week, and it also takes 30 min to measure continuously
  systolic and diastolic pressure are measured at rest, during hospital-based physical training.
Perceived dyspnea | It takes less than one minute to evaluate perceived dyspnea.
  Rating of perceived dyspnea is measured by using Borg scale at rest, during hospital-based physical training, and home-based physical activity. The most widely used tool is the "Borg scale", with rating ranges from 0 (nothing at all) to 10 (extremely dyspnea).
Oxygen saturation | Hospital-based physical training takes 30 minutes, once a week, and it also takes 30 min to measure continuously
  Oxygen saturation is continuously monitored by pulse oximetry throughout Hospital-based physical training.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Ying Wang, Phd, Study Chair — National Taiwan University
Locations (1):
- Physical Therapy Center at National Taiwan University Hospital, Taipei, Taiwan